CLINICAL TRIAL: NCT00046397
Title: A Phase I/II Clinical Trial of Modified Vaccinia Virus Ankara (MVA) to Evaluate Its Safety, Dosing Schedule, Immunogenicity and Protective Efficacy Against Dryvax Challenge in Vaccinia-Naive Individuals
Brief Title: Phase I Trial of Smallpox Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 020316; 02-I-0316
Record Dates: First submitted 2002-09-27; First posted 2002-09-30 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-08

CONDITIONS: Healthy
Keywords: Smallpox; Vaccine; Vaccination; Variola; Adults; Smallpox Vaccine; Healthy Volunteer; Small Pox
MeSH Terms: conditions — Smallpox

INTERVENTIONS:
Drug: Modified Vaccinia Virus Ankara TBC-M

SUMMARY:
This study will test the safety of an experimental vaccine called Modified Vaccinia Virus Ankara (MVA) for use against the smallpox virus. It will also investigate how many injections of MVA are needed to produce immunity against vaccinia virus, which is closely related to the smallpox virus. An effective smallpox vaccine exists, but it can cause side effects that, on rare occasions, can be life-threatening. The FDA gave new license approval for Dryvax on 10/25/02, but has not been used in the general population since smallpox was eradicated worldwide. Both the MVA and Dryvax® (Registered Trademark) vaccines are made using the vaccinia virus, however the MVA vaccine contains a more attenuated, or weakened, form of the virus. [http://www.fda.gov/cber/products/smalwye102502.htm]

Healthy normal volunteers between 18 and 30 years of age, who have never been vaccinated with a smallpox vaccine, may be eligible for this study. Candidates will be screened with a medical history, physical examination, and blood and urine tests, including an HIV test and a pregnancy test for women of childbearing potential.

MVA, placebo and Dryvax® (Registered Trademark) will be administered by different methods. The MVA vaccine and placebo are injected into an arm muscle with a needle and syringe. The Dryvax® (Registered Trademark) vaccine is administered, as it was for many years, with a special forked needle that is poked lightly into the skin of the upper arm, usually 15 times, in a process called scarification. When the vaccine works, a small pus-filled blister forms, followed by a scab and then scarring at the site of the vaccination. The formation of the blister and scab is called a take, indicating that the vaccine is effective and is evidence of the development of immunity. The development of a take suggests that an individual will be protected against smallpox for at least a few years. If scarification does not take, it can either mean that the person already has immunity or that the vaccine did not work.

Participants will be assigned to groups, as well as, product randomly. For instance, the first study participant could be enrolled into group 3. The Dryvax® (Registered Trademark) dose is given as a challenge to see if the person has a take. A reduced take response or no take, could suggest that MVA is able to produce an immune response. The dosing schedules vary from 12 to 24 weeks and volunteers are in the study a total of 24 to 36 weeks, depending on the number of injections.

Participants will be observed for at least 1 hour after each injection. They will come to the clinic a week after MVA or placebo injections and at least twice a week after Dryvax® (Registered Trademark) for about 21 days to have the injection site evaluated and photographed. At each visit, participants will be asked about how they are feeling and if they are taking any medications. Blood and urine tests will be done on injection days and at follow up visits scheduled 1 and 4 weeks after each immunization as well as 12 weeks after the Dryvax® (Registered Trademark) challenge dose. Additional tests may be done between visits if medically necessary.

DETAILED DESCRIPTION:
Phase I/II, randomized, placebo-controlled, double-blinded, schedule finding study of MVA. The hypothesis is that MVA will be safe in humans when administered by intramuscular (IM) injection and will result in an immune response comparable to that observed after Dryvax primary vaccination. The primary objectives include: evaluating the safety of MVA administered by intramuscular (IM) injection on single and multidose schedules and identifying a schedule of MVA that provides clinical evidence of protection against vaccinia (Dryvax) challenge. The secondary objectives are to compare the immunogenicity of Dryvax and MVA as measured by vaccinia-specific neutralizing antibody, ELISA, and intracellular cytokines assays and by a variola-specific neutralizing antibody assay that will be conducted at the CDC on a subset of samples.

ELIGIBILITY:
INCLUSION CRITERIA:

A participant must meet all of the inclusion criteria, as follows:

Age: at least 18 years and birth year no earlier than 1964.

Available for follow-up for the duration of the study (maximum of 28 weeks; varies according to schedule).

Able and willing to sign the informed consent form.

Willing to have blood samples that will be stored for future research.

In good general health, without clinically significant medical history, physical examination findings or laboratory results.

Hematocrit greater than or equal to 34 percent for women; greater than or equal to 38 percent for men.

White cell count within institutional normal limits.

Differential either within institutional normal range or accompanied by site physician approval.

Total lymphocyte count greater than of equal to 1000 cells/mm3.

Absolute CD4 count greater than or equal to 400 cells/mm3.

Platelets within institutional normal limits.

ALT (SGPT) less than or equal to institutional upper normal limit.

Serum creatinine less than or equal to 1.3 mg/dL and calculated creatinine clearance (CrCl) greater than or equal to 55 mL/min using the formula below:

* Male CrCl (mL/min) &eq; 140 - age (yrs)] x [body wt (kg)] divided by 72 x [serum Cr (mg/dL)]
* Female CrCl (mL/min) &eq; [140 - age (yrs)] x [body wt (kg) x 0.85] divided by 72 x [serum Cr (mg/dL)]

Normal urinalysis defined as: negative glucose, negative or trace protein, and negative or trace hemoglobin.

Negative hepatitis B surface antigen (HBsAg).

Negative anti-HCV or negative HCV PCR if the anti-HCV is positive.

Negative HIV ELISA and HIV PCR (volunteers who have previously participated in an HIV vaccine study are eligible with positive ELISA if western blot is indeterminate or negative and HIV PCR is negative).

Negative Beta-HCG serum pregnancy test for women presumed to be of reproductive potential.

A female participant must meet one of the following criteria: a) no reproductive potential due to menopause (one year without menses), hysterectomy, bilateral oophorectomy, or tubal ligation; b) agrees to consistently practice contraception at least 30 days prior to enrollment and throughout the duration of the study by means of IUD, hormone-based therapy (e.g., contraceptive pills, Norplant or Depo-Provera or other FDA-licensed methods).

Able to provide proof of identity to the acceptance of the study clinician completing the enrollment process.

EXCLUSION CRITERIA:

Volunteers are excluded from study participation if one or more of the following criteria applies:

Prior vaccination with any vaccinia product.

Diseases or conditions that cause immunodeficiency (examples are HIV AIDS, leukemia, lymphoma, generalized malignancy, agammaglobulinemia, history of transplantation, or therapy with alkylating agents, antimetabolites, radiation, or oral or parenteral corticosteroids).

In close physical contact (household or at work) with an individual who has the diseases or conditions that cause immunodeficiency.

History of eczema, even if the condition is mild or not presently active.

In close physical contact (household or at work) with an individual who has eczema even if mild or not presently active.

Acute or chronic skin conditions such as atopic dermatitis, burns, impetigo, or varicella zoster (shingles).

Household member who is pregnant.

Women who are breast-feeding.

Household member less than 1 year old or work with children less than 1 year old.

Serious, life-threatening allergies to antibiotics polymixin B, streptomycin, tetracycline, neomycin, or cidofovir.

Allergy to eggs or blood products (including immunoglobulin products) or hypersensitivity to probenicid or sulfa-containing medications.

Receipt of live attenuated viruses within 30 days prior to enrollment.

Receipt of subunit or killed vaccines within 14 days prior to enrollment.

Use of investigational research agents within 30 days prior to enrollment.

Receipt of blood products within 120 days prior to HIV screening.

Receipt of immunoglobulin within 60 days prior to HIV screening.

History of serious adverse reactions to vaccines such as anaphylaxis or related symptoms such as hives, respiratory difficulty, angioedema and abdominal pain.

History of type I or type II diabetes mellitus except gestational diabetes or diabetes controlled with diet alone.

Participant currently taking anti-TB prophylaxis or therapy.

History of seizure disorder other than: 1) febrile seizures under the age of two, or 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) a singular seizure more than 3 years ago.

Bleeding disorder diagnosed by a physician (e.g., factor deficiency, coagulopathy, or platelet disorder that requires special precautions).

Splenectomy

Hypertension that is not well controlled by medication or is more than 150/100 at enrollment.

Psychiatric condition that precludes compliance with the protocol; past or present psychoses; past or present bipolar disorder requiring therapy that has not been well-controlled on medication within the past two years; disorder requiring lithium; suicidal ideation within the five years prior to enrollment.

Any medical, psychiatric, social condition, or occupational or other responsibility that, in the judgment of the investigator, would interfere with or serve as a contraindication to adherence to the study protocol or ability to give informed consent.

History of military service 1989 or earlier.

History of cardiomyopathy, myocardial infarction, angina, congestive heart failure, coronary artery disease, stroke, transient ischemic attack or history of 3 or more risk factors for coronary heart disease from the following list:

current cigarette smoking;

high blood pressure diagnosed by a doctor;

high blood cholesterol diagnosed by a doctor;

diabetes diagnosed by a doctor;

a first degree relative (father, mother, brother, sister) who had coronary artery disease before the age of 50.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 195
Dates: Start 2002-09; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

REFERENCES:
- [Background] Stittelaar KJ, Osterhaus AD. MVA: a cuckoo in the vaccine nest? Vaccine. 2001 Jun 14;19(27):V-VI. doi: 10.1016/s0264-410x(01)00171-2. No abstract available. PMID 11395217
- [Background] Henderson DA, Inglesby TV, Bartlett JG, Ascher MS, Eitzen E, Jahrling PB, Hauer J, Layton M, McDade J, Osterholm MT, O'Toole T, Parker G, Perl T, Russell PK, Tonat K. Smallpox as a biological weapon: medical and public health management. Working Group on Civilian Biodefense. JAMA. 1999 Jun 9;281(22):2127-37. doi: 10.1001/jama.281.22.2127. PMID 10367824
- [Background] Henderson DA. The looming threat of bioterrorism. Science. 1999 Feb 26;283(5406):1279-82. doi: 10.1126/science.283.5406.1279. PMID 10037590